CLINICAL TRIAL: NCT00588276
Title: Pilot Evaluation of 124I-Iodo-Azomycin Galacto-Pyranoside (*IAZGP) Positron Emission Tomography (PET) in the Imaging of Hypoxic Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 05-023
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Cervical Cancer; HEENT Cancer; Renal Cancer; Uterine Cancer; CERVIX UTERI NOS; RECTUM
Keywords: measurable disease; locally advanced disease
MeSH Terms: conditions — Uterine Cervical Neoplasms; Kidney Neoplasms; Uterine Neoplasms

ARMS (1):
- 1 (Experimental): Patients will receive 124IAZGP(124I-Iodo-Azomycin Galacto-Pyranoside).
  Interventions: Radiation: 124I-Iodo-Azomycin Galacto-Pyranoside

INTERVENTIONS:
Radiation: 124I-Iodo-Azomycin Galacto-Pyranoside — You will receive the radioactive tracer through an injection in your vein. Blood (about 5 tablespoons in all) will be taken after the radioactive tracer has been given. Over the course of study day 1, bloods will be drawn 8 times and then 4 more times on study day 2. You will undergo three *IAZGP PET scans, one shortly after you receive the injection, one later the same day and one the following day. Each scan will take about an hour. This means you would be asked to come back 2 days in a row.

SUMMARY:
The purpose of this study is to evaluate low oxygen areas called hypoxia within the tumor. These low oxygen areas are thought to be the reason why tumors are more resistant to radiation treatment. A tracer is an extremely small quantity of a substance. Tracer to which radioactivity has been attached may be used to "trace" events in the body. A tracer called iodo-azomycin galactopyranoside (or *IAZGP) appears to be able to detect low oxygen areas within tumor.

Radioactive iodine in this molecule can be detected by an imaging technique called a PET scan. This present study involves obtaining three scans using this new imaging technique. The goal of carrying out many scans is to determine which scan will best show any areas in your tumor that may have low levels of oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have locally advanced cancer as determined by currently accepted diagnostic work-up, including CT/MR/US.
* KPS >70%.
* Patients must be > or equal to 18 years of age.

Exclusion Criteria:

* Patients will be excluded from the study if they fulfill any of the following criteria:
* Patients with abnormal baseline thyroid function tests, or any thyroid disorder including but not limited to hypothyroidism and thyroiditis. Patients with thyroid cancer who have had a thyroidectomy are not excluded.
* Patients who are pregnant or lactating.
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
* Patients who cannot tolerate being in the PET scanner for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To describe imaging findings in human cancer with the new hypoxia tracer 124IAZGP and PET/CT | at least once at approximately 6 hours and/or 24 hours after radiotracer administration.
To evaluate the biodistribution of 124IAZGP using serial PET imaging and to estimate blood radioactivity | 5, 15, 30 and 60 minutes after 124IAZGP, and before and after each. A 5-mL volume of blood will be drawn at each sampling time point.
To obtain further human dosimetry data with 124IAZGP | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Schöder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] O'Donoghue JA, Guillem JG, Schoder H, Lee NY, Divgi CR, Ruby JA, Humm JL, Lee-Kong SA, Burnazi EM, Cai S, Carlin SD, Leibold T, Zanzonico PB, Ling CC. Pilot study of PET imaging of 124I-iodoazomycin galactopyranoside (IAZGP), a putative hypoxia imaging agent, in patients with colorectal cancer and head and neck cancer. EJNMMI Res. 2013 Jun 3;3(1):42. doi: 10.1186/2191-219X-3-42. PMID 23731770
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org